CLINICAL TRIAL: NCT01122134
Title: Pharmacokinetics and Pharmacodynamics of Intravenous Artesunate in Treatment of Severe Malaria in Ugandan Patients
Brief Title: Pharmacokinetics and Pharmacodynamics of Intravenous Artesunate for Severe Malaria Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Makerere University (Other)
Responsible Party: Pauline Byakika-Kibwika, INTERACT, Makerere University
Other Study IDs: CPR 07
Record Dates: First submitted 2010-05-10; First posted 2010-05-13 (Estimated); Last update posted 2010-05-13 (Estimated); Status verified 2010-05

CONDITIONS: Severe Malaria
Keywords: severe; malaria; artesunate; intravenous
MeSH Terms: conditions — Malaria; Lymphoma, Follicular

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples collected for artesunate drug assays
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 20 adults with severe malaria: 20 adult patients admitted with severe malaria
  Interventions: Drug: intravenous artesunate

INTERVENTIONS:
Drug: intravenous artesunate — Intravenous artesunate in a dose of 2.4 mg/kg at start of treatment, 2.4 mg/kg 12 hours later and 2.4 mg/kg/day until the patient is able to tolerate oral therapy. The minimum duration of IV treatment will be 24 hours.
  Other Names: Artesun®

SUMMARY:
Intravenous artesunate is highly effective with rapid schizonticidal action and improved clinical outcome

DETAILED DESCRIPTION:
The current first line treatment for severe malaria in Uganda is intravenous quinine with artemisinin derivatives as an alternative. Intravenous artesunate, a water soluble artemisinin derivative is more effective than quinine with faster schizonticidal action and improved clinical outcome. It is generally well tolerated and safe. This study aims is to assess the pharmacokinetics, pharmacodynamics and safety of IV artesunate in treatment of severe malaria in adults admitted to Mulago National Referral and Teaching hospital, Uganda.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years and above
2. With severe malaria according to the following ciriteria:
3. A positive blood smear for malaria with P. falciparum mono-infection with parasitemia > 500 parasites/ul of blood
4. Who according to the attending physician require parenteral treatment and admission for malaria
5. Willing to participate in the study
6. Who are or whose first degree parents/caretakers are able to provide written informed consent

Exclusion Criteria:

1. Patients with history of prior antimalarial use within the last 72 hours
2. Pregnant women
3. Patients with contraindications to taking the study drugs
4. Patients taking known inhibitors or inducers of cytochrome P450 -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study are patients aged 18 years and above. The accessible population will be patients of 18 years and above who present to Mulago hospital with severe malaria. The study population will include patients aged 18 years and above presenting with severe malaria, who fulfill study eligibility criteria and are enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-08 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameters; total area under the plasma concentration vs. time curve (AUC) of artesunate and DHA, maximum plasma concentration (Cmax), time to attain maximum concentration, elimination half life | 6 hours
  Pharmacokinetic parameters for artesunate and dihydroartemisinin

SECONDARY OUTCOMES:
Time to 50% parasite clearance (PCT50) | 7 days
  Time to 50% parasite clearance (PCT50) parasite clearance rates and clinical recovery

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Byakika-Kibwika, MSc, MMed, Principal Investigator — Makerere University
Locations (1):
- Mulago National Referral hospital, Kampala, Uganda

REFERENCES:
- [Derived] Byakika-Kibwika P, Lamorde M, Mayito J, Nabukeera L, Mayanja-Kizza H, Katabira E, Hanpithakpong W, Obua C, Pakker N, Lindegardh N, Tarning J, de Vries PJ, Merry C. Pharmacokinetics and pharmacodynamics of intravenous artesunate during severe malaria treatment in Ugandan adults. Malar J. 2012 Apr 27;11:132. doi: 10.1186/1475-2875-11-132. PMID 22540954